CLINICAL TRIAL: NCT01310036
Title: An Open-Label Multicenter Study of Erlotinib (Tarceva®) as First Line Therapy Until and Beyond RECIST Progression in NSCLC Patients Who Harbour EGFR Mutations
Brief Title: A Study of Tarceva (Erlotinib) as First Line Therapy in Participants With Non-Small Cell Lung Cancer Harbouring Epidermal Growth Factor Receptor (EGFR) Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25637
Record Dates: First submitted 2011-02-18; First posted 2011-03-07 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (1):
- Erlotinib (Experimental): Erlotinib 150 mg daily
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg was administered orally daily until disease progression or unacceptable toxicity.
  Other Names: Tarceva

SUMMARY:
This open-label, single arm study will evaluate the safety and efficacy of Tarceva (erlotinib) as first-line therapy in participants with stage IV or recurrent non-small cell lung cancer who harbour epidermal growth factor receptor (EGFR) mutations. All participants will receive Tarceva 150 mg daily orally until disease progression or unacceptable toxicity occurs. At the investigator's discretion, participants may receive Tarceva beyond disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Stage IV or recurrent non-small cell lung cancer (NSCLC)
* Presence of mutation(s) in exon 18 through exon 21 of epidermal growth factor receptor (EGFR), (except T790M single mutation only)
* Measurable disease (at least one lesion >= 10 mm in longest diameter)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Patients with T790M single mutation only
* Prior exposure to agents directed at the human epidermal receptor (HER) axis, e.g. erlotinib, gefitinib, cetuximab, trastuzumab
* Prior chemotherapy or systemic anti-cancer therapy for advanced NSCLC disease
* Symptomatic or uncontrolled central nervous system (CNS) metastases
* Other malignancy within the last 5 years, except for carcinoma in situ of the cervix, or basal or squamous cell carcinoma of the skin, or surgically treated localized prostate cancer, or surgically treated ductal cell carcinoma in situ of the breast
* Any significant ophthalmologic abnormality
* Pre-existing parenchymal lung disease such as pulmonary fibrosis
* Use of coumarins (for anti-coagulation therapy the use of low molecular weight heparin is recommended instead)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2011-04-30 (Actual); Primary Completion 2014-02-14 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Hong Kong (3):
  - Princess Margaret Hospital; Oncology, Hong Kong
  - Queen Elizabeth Hospital; Clinical Oncology, Hong Kong
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- South Korea (6):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gil Hospital. Gachon University, Incheon
  - Asan Medical Center; Medical Oncology, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Yonsei University Severance Hospital; Medical Oncology, Seoul
- Taiwan (10):
  - Changhua Christian Hospital; Internal Medicine, Changhua
  - Kaohsiung Chang Gung Memorial Hospital; Dept of Internal Medicine, Kaohsiung City
  - Veterans General Hospital; Internal Medicine, Kaohsiung City
  - China Medical University Hospital; Pulmonary and Critical Care Medicine, Taichung
  - Taichung Veterans General Hospital; Dept of Internal Medicine, Taichung
  - National Cheng Kung Uni Hospital; Dept of Hematology and Oncology, Tainan
  - Chi-Mei Medical Centre; Hematology & Oncology, Tainan
  - National Taiwan Uni Hospital; Internal Medicine, Taipei
  - Taipei Veterans General Hospital; Chest Dept , Section of Thoracic Oncology, Taipei
  - Chang Gung Medical Foundation - Linkou; Chest Dept, Taoyuan District
- Thailand (3):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - Pramongkutklao Hospital; Medicine - Medical Oncology Unit, Bangkok
  - Songklanagarind Hospital; Department of Internal Medicine, Division of Respiratory, Songkhla

REFERENCES:
- [Derived] Park K, Yu CJ, Kim SW, Lin MC, Sriuranpong V, Tsai CM, Lee JS, Kang JH, Chan KC, Perez-Moreno P, Button P, Ahn MJ, Mok T. First-Line Erlotinib Therapy Until and Beyond Response Evaluation Criteria in Solid Tumors Progression in Asian Patients With Epidermal Growth Factor Receptor Mutation-Positive Non-Small-Cell Lung Cancer: The ASPIRATION Study. JAMA Oncol. 2016 Mar;2(3):305-12. doi: 10.1001/jamaoncol.2015.4921. PMID 26720423

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib
Started | 208
Completed | 6
Not Completed | 202
Not completed — Administrative/other | 10
Not completed — Withdrew Consent | 11
Not completed — Refused Treatment/Did not Cooperate | 4
Not completed — Progression of Disease | 164
Not completed — Death | 1
Not completed — Adverse event or intercurrent illness | 12

BASELINE CHARACTERISTICS:
Population: Of the 208 participants who were enrolled in the study, one participant was excluded from the baseline analysis population.
Arm/Group | Erlotinib
Number analyzed (Participants) | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 78

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Per RECIST, v. 1.1 (PFS1)
Description: PFS1 was defined as time from first dose until documented progressive disease (PD), assessed per Response Evaluation Criteria in Solid Tumors RECIST, v. 1.1, or death from any cause, whichever occurred first. PD was defined as: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline; an absolute increase of at least 5 mm in the sum of diameters of target lesions; and the appearance of one or more new lesions.
Time Frame: Approximately 68 months
Population: The per protocol population included participants who had EGFR mutations confirmed by a study-designated central laboratory.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 148
months | 11.000 [9.267 to 11.200]

2. Secondary Outcome: Progression-free Survival Per Investigator (PFS2)
Description: PFS2 was defined as time from first study dose to off-erlotinib progressive disease (PD), assessed by the investigator based on overall clinical evaluation.
Time Frame: Approximately 68 months
Population: The per protocol population included participants who had EGFR mutations confirmed by a study-designated central laboratory. Data are reported for evaluable participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 69
months | 15.000 [13.067 to 18.700]

3. Secondary Outcome: Objective Response Rate (ORR) for All Participants and Participants With EGFR Mutation E19del or L858R
Description: ORR was defined as the occurrence of either a confirmed complete (CR) or a partial response (PR, as a best overall response), as determined by RECIST, v. 1.1 criteria. CR was defined as disappearance of all target lesions. PR was defined as least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Approximately 68 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 148
percentage of participants
  All Participants | 72.3 [64.3 to 79.3]
  EGFR Mutation E19del or L858R: number analyzed (Participants) | 144
  EGFR Mutation E19del or L858R | 72.9 [64.9 to 80.0]

4. Secondary Outcome: Disease Control Rate (DCR) for All Participants and Participants With EGFR Mutation E19del or L858R
Description: DCR was defined as CR + PR + Stable disease (SD). CR was defined as disappearance of all target lesions. PR was defined as least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. PD was defined as: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline; an absolute increase of at least 5 mm in the sum of diameters of target lesions; and the appearance of one or more new lesions.
Time Frame: Approximately 68 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 148
percentage of participants
  All Participants | 84.5 [77.6 to 89.9]
  EGFR Mutation E19del or L858R: number analyzed (Participants) | 144
  EGFR Mutation E19del or L858R | 85.4 [78.6 to 90.7]

5. Secondary Outcome: Progression-free Survival for Participants With EGFR Mutation E19del or L858R Per RECIST, v. 1.1 (PFS1)
Description: as for outcome 1
Time Frame: Approximately 68 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 144
months | 11.000 [9.267 to 11.200]

6. Secondary Outcome: Overall Survival (OS) for All Participants and Participants With EGFR Mutation E19del or L858R
Description: OS was defined as the time from baseline to the date of death from any cause.
Time Frame: Approximately 68 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 148
months
  All Participants | 31.633 [28.100 to 36.133]
  EGFR Mutation E19del or L858R: number analyzed (Participants) | 144
  EGFR Mutation E19del or L858R | 31.800 [28.100 to 36.133]

7. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug.
Time Frame: Approximately 68 months
Population: The safety population included all participants who received at least one dose study medication and had at least one post baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 207
participants | 206

8. Secondary Outcome: Correlation Between EGFR Mutations in Plasma and Clinical Outcome (ORR/PFS/OS)
Description: This outcome measure was not assessed.
Time Frame: Approximately 68 months
Population: Data were not collected.
Arm/Group | Erlotinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 68 months
Description: The safety population included all participants who received at least one dose study medication and had at least one post baseline safety assessment.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 59/207
Other Adverse Events (participants affected / at risk) | 206/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=207)
Pneumonia (Infections and infestations) | 10
Cellulitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Dengue fever (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Parainfluenzae virus infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal scalded skin syndrome (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Pneumoconiosis (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 2
Death (General disorders) | 2
Cerebral infarction (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Neuritis cranial (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Hepatitis (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Arthritis bacterial (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=207)
Rash (Skin and subcutaneous tissue disorders) | 110
Pruritus (Skin and subcutaneous tissue disorders) | 73
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 56
Dry skin (Skin and subcutaneous tissue disorders) | 53
Alopecia (Skin and subcutaneous tissue disorders) | 34
Acne (Skin and subcutaneous tissue disorders) | 20
Skin exfoliation (Skin and subcutaneous tissue disorders) | 13
Nail disorder (Skin and subcutaneous tissue disorders) | 14
Eczema (Skin and subcutaneous tissue disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 124
Stomatitis (Gastrointestinal disorders) | 43
Nausea (Gastrointestinal disorders) | 25
Constipation (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 23
Mouth ulceration (Gastrointestinal disorders) | 14
Abdominal pain upper (Gastrointestinal disorders) | 11
Mucosal inflammation (General disorders) | 32
Fatigue (General disorders) | 30
Chest pain (General disorders) | 19
Pyrexia (General disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 56
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 21
Productive cough (Respiratory, thoracic and mediastinal disorders) | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16
Paronychia (Infections and infestations) | 62
Conjunctivitis (Infections and infestations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 45
Hypokalaemia (Metabolism and nutrition disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 28
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Alanine aminotransferase increased (Investigations) | 28
Aspartate aminotransferase increased (Investigations) | 22
Blood bilirubin increased (Investigations) | 12
Headache (Nervous system disorders) | 25
Dizziness (Nervous system disorders) | 20
Dry eye (Eye disorders) | 25
Insomnia (Psychiatric disorders) | 19
Anaemia (Blood and lymphatic system disorders) | 17
Upper respiratory tract infection (Infections and infestations) | 11
Weight decreased (Investigations) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.